CLINICAL TRIAL: NCT07338682
Title: Evaluation of the Effect of L-Arginine on the Cognitive Function in Geriatric Patients, A Randomized Clinical Trial
Brief Title: Evaluation of the Effect of L-Arginine on the Cognitive Function in Geriatric Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German University in Cairo (Other)
Responsible Party: Principal Investigator, Rama Elmor, Teaching Assistant/Pharmacist, German University in Cairo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L-Arg_on_MCI_in_Geriatrics
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cognition Disorders in Old Age; Cognitive and Behavioral Impairment
Keywords: L-arginine; Cognitive impairment; Geriatrics; Elderly; Cognitive Function; Nitric Oxide
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Arginine

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-Arginine (Experimental): 6 grams sachets of L-arginine once daily
  Interventions: Dietary Supplement: L-Arginine
- Placebo (Placebo Comparator): Matching placebo once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-Arginine — 6 grams L-arginine sachets taken orally once daily
  Arms: L-Arginine
Other: Placebo — Matching Placebo of L-arginine
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effect of L-arginine supplementation on cognitive function in geriatric patients. Eligible participants will receive either L-arginine (6 grams once daily) or placebo, and their cognitive performance will be assessed using validated cognitive assessment tools over the study period. The participants will receive the intervention for 4 weeks and followed up every 2 weeks. The primary outcome is improvement in cognitive function, while secondary outcomes include safety, tolerability, and quality of life measures. The findings may provide evidence for the potential role of L-arginine in supporting cognitive health in elderly populations.

DETAILED DESCRIPTION:
Cognitive decline is a common problem in the geriatric population and can significantly affect independence, quality of life, and overall health outcomes. Emerging evidence suggests that L-arginine, a semi-essential amino acid and precursor for nitric oxide synthesis, may play a role in improving cerebral blood flow and neuronal function. These mechanisms could potentially contribute to better cognitive performance in elderly individuals.

This study is designed to evaluate the effect of L-arginine supplementation on cognitive function in geriatric patients. Participants who meet eligibility criteria will be randomized to receive either L-arginine supplementation or placebo. Cognitive function will be assessed at baseline and at defined intervals during the study period using validated neurocognitive assessment tools. Additional measures will include safety monitoring, tolerability, and secondary assessments such as quality of life indices.

The primary objective is to determine whether L-arginine supplementation improves cognitive function. Secondary objectives include evaluating the anti-inflammatory, antioxidant effect and safety profile of L-arginine in older adults and assessing its potential impact on daily living and overall well-being. The results of this study may provide valuable insights into the role of L-arginine in supporting cognitive health in elderly populations and inform future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age >60 years
* Montreal Cognitive Assessment (MoCA) test score from 10-25 (mild to moderate cognitive impairment)

Exclusion Criteria:

* Presence of neurodegenerative diseases (e.g.: Alzheimer's disease, Parkinson's disease, Huntington's disease, Multiple Sclerosis)
* Patients with history of L-arginine intolerance or allergy
* Patients with asthma
* Patients who recently had an acute myocardial infarction
* Patients with history of stroke within 1 yaear
* Patients who started or discontinued medications that may affect cognitive function (e.g., CNS psychotropics, antihistamines, or acetylcholinesterase inhibitors) during the study period.
* Patients who initiated or stopped antihypertensive medications during the study period.
* Patients who initiated or stopped antidiabetic medications during the study period.
* Patients who initiated or stopped antihyperlipidemic medications during the study period.
* Patients prescribed medications for depression, anxiety, or stress that may impact cognitive function
* Patients on nitrates, phosphodiesterase-5 inhibitors, potassium sparing diuretics
* Refusal to provide written informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | at baseline, after 2 weeks, and after 4 weeks
  MOCA is a is a brief cognitive screening tool used to detect mild cognitive impairment (MCI) and early dementia. It assesses multiple cognitive domains including memory, attention, executive function, language, visuospatial skills, abstraction, calculation, and orientation. The score ranges from 0- 30. The higher the score the better the cognition. The normal range is from 26-30.

SECONDARY OUTCOMES:
Depression, Anxiety, Stress Scales-21 (DASS-21) | at baseline, after 2 weeks, and after 4 weeks
  DASS-21 is a short self-report questionnaire used to assess depression, anxiety, and stress over the past week. It consists of 21 items, with 7 items for each subscale, rated on a 4-point Likert scale. Each subscale has a raw score range of 0-21and the higher the score the worse the outcome of symptoms of depression, anxiety, or stress.
The World Health Organization Quality of Life (WHOQOL-BREF) | at baseline, after 2 weeks, and after 4 weeks
  WHOQOL-BREF is a brief, self-administered questionnaire that assesses an individual's perceived quality of life. It consists of 26 items covering four domains: physical health, psychological health, social relationships, and environment. Score can range from 0-100 for each domain with higher scores meaning a better quality of life.
ADMA | at baseline and after 4 weeks
  Asymmetric dimethylarginine
MDA | at baseline and after 4 weeks
  Malondialdehyde
CRP | at baseline and after 4 weeks
  C-reactive protein
Lipid Profile | at baseline and after 4 weeks
Kidney Function test | at baseline and after 4 weeks
  Serum Creatinine
Liver Function Tests | at baseline and after 4 weeks
  ALT and AST

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Department, Al-Azhar University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No